CLINICAL TRIAL: NCT03539016
Title: Epidemiological Study on Clinical Features of Chronic Hepatitis B Virus Infection During Pregnancy and Hepatitis B Virus Mother-to-child Transmission (Shield Study Phase Ⅰ)
Brief Title: Observational Study on Pregnant Women With Chronic Hepatitis B and Their Infants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: SHIELD-01
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B, Mother-to-child transmission
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study was conducted to observe the clinical features during pregnancy in women with chronic hepatitis B virus infection and mother-to-child transmission of hepatitis B virus.

ELIGIBILITY:
Inclusion Criteria:

1. Gestation of 4-32 weeks
2. HBsAg+ > 6 months, HBeAg+/-
3. Informed consent signed voluntarily
4. Good compliance and able to be followed up as planned

Exclusion Criteria:

1. Coinfection with hepatitis C virus or human immunodeficiency virus;
2. Comorbidities of other severe conditions that hinder compliance with follow ups and because of that, the subjects are anticipated to be unable to complete the project.;
3. Unable or unwilling to use mobile health tools.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant woman
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Rate of mother-to-child transmission | Infants from 7 to 12 months of age
Rate of hepatitis flare during pregnancy and postpartum | up to postpartum weeks 6-8

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Nanfang Hospital, Guangzhou, Guangdong
  - 302 military hospital of China, Beijing
  - Beijing YouAn Hospital, Beijing
  - Fifth Affiliated Hospital of Southern Medical University, Guangzhou
  - Guangzhou No. 8 People's Hospital, Guangzhou
  - Third Affiliated Hospital of Southern Medical University, Guangzhou
  - Zhujiang Hospital, Guangzhou
  - Jiujiang Maternal and Child Care Service Centre, Jiujiang
  - Third Hospital of Jiujiang, Jiujiang
  - Second Hospital of Nanjing, Nanjing

IPD SHARING:
Plan to Share IPD: Undecided